CLINICAL TRIAL: NCT01443195
Title: Iron Metabolism in Small Pre Term Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B and Pediatric Hematology Unit, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0035-11-EMC
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Preterm; Iron Metabolism; Iron Overload
MeSH Terms: conditions — Premature Birth; Iron Overload | interventions — Iron, Dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron suplementation (Experimental): Iron supplementation with IPC in a dose of 4 mg/kg/day of elemental iron started not before 4 weeks of age and as soon as 120 ml/kg/day of enteral feedings is tolerated given together with the first morning meal
  Interventions: Drug: Iron preparation

INTERVENTIONS:
Drug: Iron preparation — Iron supplementation with IPC in a dose of 4 mg/kg/day of elemental iron started not before 4 weeks of age and as soon as 120 ml/kg/day of enteral feedings is tolerated given together with the first morning meal. Serum samples will be obtained at 3 different times:
  1. Before starting iron supplementation (maximum one week before).
  2. At the beginning of iron supplementation in order to assess early signs of erythropoiesis, iron overload or free iron (day 4 - 7 days of supplementation).
  3. Before discharge from hospitalization in order to asses the iron metabolism and sings of iron deficiency (At least more than 2 weeks of supplementation).

SUMMARY:
Iron is an essential micronutrient that plays an important role in cellular functions of all microorganisms. Both iron deficiency and iron excess during the early weeks of life can have severe effects on neurodevelopment that may persist into adulthood and may not be corrected by restoration of normal iron levels.

Iron overload remains a significant concern in preterm infants because they have low levels of iron-binding proteins and immature antioxidant systems.

The aim of the study is to evaluate if iron supplementation is required/necessary in VLBW Very Low Birth Weight (less than 1500 grams) and to assess the efficacy and safety of the iron supplementation practice for VLBW preterm infants as implemented in the Neonatal Intensive Care Unit (NICU) at the Ha'Emek Medical Center, Afula, Israel.

DETAILED DESCRIPTION:
Primary objectives

1. The aim of the study is to investigate the presence and level of Cryptic LPI in pre term infants plasma before and during enteral iron supplementation.
2. To assess the iron status in preterm infants and correlated them with clinical parameters: the blood transfusions given and the amount of blood obtained for routine laboratory analysis, and amount of daily iron intake through diet (human milk or formula)
3. To identify which preterm infants are at risk for iron deficiency or iron overload.
4. To investigate laboratory tests, Hepcidin and CHr, for the assessment of iron metabolism in preterm infants.

Secondary objectives To review the current guidelines in use for monitoring iron status and prevention of iron deficiency in VLWP.

To implement future new guidelines for monitoring iron therapy and iron supplementation in pre terms infants if the results suggest changes in the current policy.

Treatment guidelines:

Erythropoietin will not be administrated. Restrictive red cell transfusion guidelines will be followed. All the premature infants included in the study will receive Vitamin E supplementation as the currently used in the NICU ward.

Iron supplementation with IPC in a dose of 4 mg/kg/day of elemental iron started not before 4 weeks of age and as soon as 120 ml/kg/day of enteral feedings is tolerated given together with the first morning meal

Patients and Methods Study population: all newborn infants VLBW and or borne at 30 weeks or less of gestational age admitted at the Ha'Emek Medical Center, NICU will be screened for study eligibility. The estimate number of patients that will be included in the study is 50 during a period of one year

Inclusion criteria:

VLBW and / or borne at 30 weeks or less of gestational age that are scheduled to receive enteral iron supplementation as part of the standard protocol currently used by the NICU. Birth weight will be not an inclusion or exclusion criteria for preterms born at 30 weeks or less.

Exclusion criteria: Major physical anomalies, renal or cardiac diseases, newborns that underwent major surgery during the study period, acute or chronic fetal blood loss, hemolytic anemia, refusal to receive parental consent.

Laboratory analyses:

Complete blood count including reticulocyte count and CHr. Serum iron, Transferrin, C Reactive Protein (CRP), erythropoietin, ferritin Serum Hepcidin and serum Cryptic LPI.

The blood samples will be obtained 3 hs after oral iron administration. The blood tests will be collected at same time of necessary routine blood tests.

The serum will be collected at last 72 hs apart of clinical events: sepsis, NEC Necrotizing Enterocolitis, Intra ventricular hemorrhage, severe illness and or blood transfusions.

Complete blood count including reticulocyte count and CHr (0.5 cc of blood in EDTA), will be performed on a cell counter at Ha'Emek Medical Center laboratory.

Serum laboratory analyses 2.5 cc of blood will be centrifuged (no more than 2 h after extraction) 0.25 cc of serum will be conserved at -700 C for the hepcidin analysis, 1 cc of serum will be conserved at -700 C for the Cryptic LPI analysis.

Serum iron, Transferrin, C Reactive Protein (CRP), erythropoietin and ferritin analysis will be performed at Ha'Emek Medical Center laboratory in the day of blood extraction immediately after blood centrifugation ( 0.5 cc of serum).

Iron saturation will be calculated from serum iron and transferrin results. Serum hepcidin will be measured by ELISA using the kit EIA-4705, DRG Instruments GmbH, Germany, Frauenbergstr at Ha'Emek Medical Center laboratory following the kit instructions.

Serum Cryptic LPI will measured by Aferrix Ltd, Rehovot, Israel.

Serum samples will be obtained at 3 different times:

1. Before starting iron supplementation (maximum one week before).
2. At the beginning of iron supplementation in order to assess early signs of erythropoiesis, iron overload or free iron (day 4 - 7 days of supplementation).
3. Before discharge from hospitalization in order to asses the iron metabolism and sings of iron deficiency (At least more than 2 weeks of supplementation).

Demographic and perinatal data will be collected, the data will include:

Ethnic origin, gender, gestational age, birth weight, Apgar score, adverse events during the neonatal period including mechanical ventilation, infections, antibiotic therapy and jaundice.

Number and amount of blood transfusions, Amount of blood obtained for routine analysis calculated by the number of blood tests.

Time of introduction of enteral feeding, kind and daily amount of human milk or formula, and amount of daily iron intake through diet.

Time of iron supplementation, dose change, days without iron supplementation will be summarized. Accumulative amount of iron supplemented till discharge, calculated by mean iron supplementation per day and per grams of weight gain will also summarized.

Follow-up of weight gain. Perinatal morbidity, and complications. Adverse reactions related to iron treatment: skin rash, vomiting, bloody stools and NEC.

Maternal last red blood count before admission for delivery will be recorded. Maternal iron, transferrin, ferritin level and Hb electrophoresis if present in maternal records,

ELIGIBILITY:
Inclusion Criteria:

* Very Low Birth Weight and / or borne at 30 weeks or less of gestational age that are scheduled to receive enteral iron supplementation as part of the standard protocol currently used by the Neonatal Intensive Care Unit.
* Birth weight will be not an inclusion or exclusion criteria for preterms born at 30 weeks or less.

Exclusion Criteria:

* Major physical anomalies,
* renal or cardiac diseases,
* newborns that underwent major surgery during the study period,
* acute or chronic fetal blood loss,
* hemolytic anemia,
* refusal to receive parental consent.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of iron status in preterm infants and identify which preterm infants are at risk for iron deficiency or iron overload. | One year
  Assessment of the iron status in preterm infants and correlated them with clinical parameters: the blood transfusions given and the amount of blood obtained for routine laboratory analysis, and amount of daily iron intake through diet (human milk or formula)and identify which preterm infants are at risk for iron deficiency or iron overload.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel